CLINICAL TRIAL: NCT03584009
Title: A Phase II, Multicenter, Randomized Study To Compare The Efficacy Of Venetoclax Plus Fulvestrant Versus Fulvestrant In Women With Estrogen Receptor-Positive, Her2-Negative Locally Advanced Or Metastatic Breast Cancer Who Experienced Disease Recurrence Or Progression During Or After CDK4/6 Inhibitor Therapy
Brief Title: A Phase II Study Comparing The Efficacy Of Venetoclax + Fulvestrant Vs. Fulvestrant In Women With Estrogen Receptor-Positive, Her2-Negative Locally Advanced Or Metastatic Breast Cancer Who Experienced Disease Recurrence Or Progression During Or After CDK4/6 Inhibitor Therapy
Acronym: Veronica
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision, no safety concerns.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO40181; 2017-005118-74 (EudraCT Number)
Record Dates: First submitted 2018-06-25; First posted 2018-07-12 (Actual); Results first posted 2021-09-27 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Estrogen Receptor-positive (ER+)/Human Epidermal Growth Factor Receptor (HER2)-Negative Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — venetoclax; Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Venetoclax + Fulvestrant (Experimental): Participants were administered Venetoclax 800mg orally once daily (QD) and Fulvestrant 500mg intramuscularly (IM) on Day 1 and 15 of Cycle 1 and Day 1 of subsequent cycles (Cycle length = 28 days).
  Interventions: Drug: Venetoclax; Drug: Fulvestrant
- Fulvestrant (Active Comparator): Participants were administered Fulvestrant 500mg only IM on Day 1 and 15 of Cycle 1 and Day 1 of subsequent cycles (Cycle length = 28 days).
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Venetoclax — Venetoclax was administered orally, 800-mg tablet beginning on Cycle 1 Day 1 until the 9th October 2020.
  Arms: Venetoclax + Fulvestrant
Drug: Fulvestrant — Fulvestrant was administered orally, 500 mg administered as two 250-mg IM injections on Cycle 1 Days 1 and 15 and on Day 1 of each subsequent 28-day cycle

SUMMARY:
This is a Phase II, multicenter, open-label, randomized study to compare the efficacy of venetoclax in combination with fulvestrant compared with fulvestrant alone in women with ER+, HER2-negative, locally advanced or Metastatic Breast Cancer (MBC) who experienced disease recurrence or progression during or after treatment with CDK4/6i therapy for at least 8 weeks. As of 9th October 2020, participants in the Venetoclax + Fulvestrant arm, have all discontinued Venetoclax treatment and have continued on Fulvestrant treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of estrogen receptor-positive (ER+) invasive carcinoma of the breast. ER+, HER2- negative invasive carcinoma of the breast with evaluable sample for BCL-2 IHC value at the time of screening. Participants who were originally diagnosed with HER2-positive breast cancer that converted to HER2-negative MBC are not eligible.
* Evidence of metastatic or locally advanced disease not amenable to surgical or local therapy with curative intent.
* Be postmenopausal or pre- or perimenopausal women amenable to being treated with the luteinizing hormone-releasing hormone (LHRH) agonist goserelin.
* Participants must not have received more than two prior lines of hormonal therapy in the locally advanced or metastatic setting. In addition, at least one line of treatment must be a CDK4/6i AND participants must have experienced disease recurrence or progression during or after CDK4/6i therapy, which must have been administered for a minimum of 8 weeks prior to progression.
* Participants for whom endocrine therapy (e.g., fulvestrant) is recommended and treatment with cytotoxic chemotherapy is not indicated at the time of entry into the study, as per national or local treatment guidelines.
* Women of childbearing potential (i.e., not postmenopausal for at least 12 months or surgically sterile) must have had a negative serum pregnancy test result at screening, within 14 days prior to the first study drug administration.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use non-hormonal contraceptive methods with a failure rate of <1% per year during the treatment period and for up to 2 years after the last dose of study drug (or based on the local prescribing information for fulvestrant). Women must refrain from donating eggs during this same period.
* Willing to provide tumor biopsy sample.
* Had at least one measurable lesion via RECIST v1.1.
* Had an Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-1.
* Had adequate organ and marrow function.
* Had a life expectancy > 3 months.
* To full fill the coagulation requirements for patient with or without therapeutic anticoagulation.

Exclusion criteria:

* Prior treatment with fulvestrant or other selective estrogen receptor degraders (SERDs), venetoclax, or any agent whose mechanism of action is to inhibit BCL-2.
* Pregnant, lactating, or intending to become pregnant during the study.
* Known untreated or active Central Nervous System (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control.
* Prior chemotherapy in the locally advanced or metastatic setting regardless of the duration of the treatment.
* Any anti-cancer therapy received within 21 days of the first dose of study drug, including chemotherapy, radiotherapy, hormonal therapy, immunotherapy, antineoplastic vaccines, or other investigational therapy. (Radiotherapy with palliative intent to non-target sites is allowed).
* Concurrent radiotherapy to any site or prior radiotherapy within 21 days of Cycle 1 Day 1 or previous radiotherapy to the target lesion sites (the sites that are to be followed for determination of a response) or prior radiotherapy to > 25% of bone marrow.
* Current severe, uncontrolled, systemic disease (e.g., clinically significant cardiovascular, pulmonary, metabolic or infectious disease.
* Any major surgery within 28 days of the first dose of study drug or anticipation of the need for major surgery during the course of study treatment.
* Consumption of one or more of the following within 3 days prior to the first dose of study drug: Grapefruit or grapefruit products; Seville oranges including marmalade containing Seville oranges; Star fruit (carambola).
* Administration within 7 days prior first dose of study treatment of Steroid therapy for anti-neoplastic intent, Strong or moderate CYP3A inhibitors or Strong or moderate CYP3A inducers.
* Need for current chronic corticosteroid therapy (> 10 mg of prednisone per day or an equivalent dose of other anti-inflammatory corticosteroids).
* Known infection with (human immunodeficiency virus) HIV or human T-cell leukemia virus 1.
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1 Day).
* Positive test results for hepatitis B core antibody (HBcAb) or hepatitis C virus (HCV) antibody at screening. Participants who were positive for HCV antibody should have been negative for HCV by PCR to be eligible for study participation. Participants with a past or resolved hepatitis B virus (HBV) infection (defined as having a positive total HBcAb and negative hepatitis B surface antigen [HbsAg]) may be included if HBV DNA is undetectable. These participants should have been willing to undergo monthly DNA testing.
* Participants who had a positive HCV antibody test are eligible for the study if a PCR assay is negative for HCV RNA.
* History of other malignancies within the past 5 years except for treated skin basal cell carcinoma, squamous cell carcinoma, non-malignant melanoma <= 1.0 mm without ulceration, localized thyroid cancer, or cervical carcinoma in-situ.
* Administration of a live, attenuated vaccine within 4 weeks prior to initiation of study treatment or anticipation of need for such a vaccine during the study.
* Cardiopulmonary dysfunction.
* Other medical or psychiatric conditions that, in the opinion of the investigatory, may interfere with the participant's participation in the study.
* Inability or unwillingness to swallow pills or receive intramuscular (IM) injections.
* History of malabsorption syndrome or other condition that would interfere with enteral absorption.
* History of inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis) or active bowel inflammation (e.g., diverticulitis).
* Concurrent hormone replacement therapy.
* Inability to comply with study and follow-up procedures.
* History or active cardiopulmonary dysfunction.
* Known hypersensitivity to any of the study medications (fulvestrant, venetoclax) or to any of the excipients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female and >= 18 years of age at time of signing Informed Consent Form
Enrollment: 103 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2021-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (40):
- United States (21):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - UC San Deigo Moores Cancer Center, La Jolla, California
  - Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - St. Joseph Health Medical Group - Annadel Medical Group, Santa Rosa, California
  - Sylvester Comprehensive Cent., Miami, Florida
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Kaiser Permanente - Moanalua Medical Center, Honolulu, Hawaii
  - Ashland-Bellefonte Cancer Center, Ashland, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital., Boston, Massachusetts
  - Mass General/North Shore Cancer, Peabody, Massachusetts
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Nebraska Hematology Onco, PC, Lincoln, Nebraska
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Cleveland Clinic, Cleveland, Ohio
  - Sanford Health System, Sioux Falls, South Dakota
  - The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - The Center for Cancer and Blood Disorders - Fort Worth, Fort Worth, Texas
  - Millennium Research & Clinical Development, Houston, Texas
  - Providence Regional Cancer Partnership, Everett, Washington
- Australia (3):
  - Mater Hospital; Patricia Ritchie Centre for Cancer Care and Research, North Sydney, New South Wales
  - Mater Misericordiae Limited, South Brisbane, Queensland
  - Peter MacCallum Cancer Center, North Melbourne, Victoria
- Canada (4):
  - Southlake Regional Health Center, Newmarket, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke - Hopital Fleurimont, Sherbrooke, Quebec
- Germany (7):
  - Hämato-Onkologische Schwerpunktpraxis am Klinikum Aschaffenburg, Aschaffenburg
  - Universitätsklinikum Erlangen; Frauenklinik, Erlangen
  - Klinikum Frankfurt Höchst GmbH, Frankfurt
  - Facharztzentrum Eppendorf, Studien GbR, Hamburg
  - Rotkreuzklinikum München; Frauenklinik, München
  - Gemeinschaftspraxis für Hämatologie und Onkologie GbR; Dechow & Decker & Nonnenbroich, Ravensburg
  - Klinikum Südstadt Rostock, Rostock
- United Kingdom (5):
  - Royal United Hospital Bath NHS Trust, Bath
  - Royal Sussex County Hospital, Brighton
  - Barts Health NHS Trust - St Bartholomew's Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 38 centers in 5 countries.
Pre-assignment Details: A total of 103 participants were randomized in this study. Of these, 101 participants received at least one dose of any study drug.
Period: Overall Study
Arm/Group | Venetoclax + Fulvestrant | Fulvestrant
Started | 51 | 52
Completed | 0 | 0
Not Completed | 51 | 52
Not completed — Death | 25 | 18
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Study Terminated by Sponsor | 22 | 30
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) population included all randomized participants whether or not they were assigned to the arm where the study treatment was administered.
Groups:
- Venetoclax + Fulvestrant: Participants were administered Venetoclax 800mg orally QD and Fulvestrant 500mg IM on Day 1 and 15 of Cycle 1 and Day 1 of subsequent cycles (Cycle length = 28 days).
- Total: Total of all reporting groups
Arm/Group | Venetoclax + Fulvestrant | Fulvestrant | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (10.6) | 58.8 (11.7) | 58.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 52 | 103
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 47 | 46 | 93
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 40 | 46 | 86
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Defined as Complete Response (CR), Partial Response (PR) or Stable Disease (SD) Lasting >= 24 Weeks, as Determined by the Investigator According to RECIST v1.1
Description: Clinical Benefit was defined as CR, PR, or SD lasting more than equal to 24 weeks from randomization in participants with measurable disease at baseline, as determined by the investigator according to Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1. Per RECIST v1.1 for target lesions assessed by CT or MRI: CR, Disappearance of all target lesions; PR, PR >= 30% decrease in the sum of diameters of target lesions (TL) taking as reference the baseline sum of diameters; SD, neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Disease Progression (PD), PD>= 20% increase in the sum of diameters of TL taking as reference the smallest sum on study(Nadir). In addition to the relative increase of 20% sum must have demonstrate an absolute increase of at least 5mm.
Time Frame: Randomization through till 6 months after the last participant is enrolled into the study (up to approximately 23 months)
Population: The Baseline Measurable Disease Population represented all randomized participants with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Venetoclax + Fulvestrant | Fulvestrant
Number analyzed (Participants) | 51 | 51
Percentage of Participants | 11.8 [4.44 to 23.87] | 13.7 [5.70 to 26.26]
Statistical Analysis 1: Comparison: Venetoclax + Fulvestrant vs Fulvestrant; Test type: Superiority; p = 0.7286, Cochran-Mantel-Haenszel — P-value is based on Stratified Analysis (Stratified by BCL2 status (High vs Low) and Lines of Therapy (2 vs 1)); Risk Difference (RD) = -1.96, 95% CI 2-sided [-16.86 to 12.94]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first occurrence of disease progression (as determined by the investigator according to RECIST v1.1) or death from any cause, whichever occurs first.
Time Frame: as for outcome 1
Population: ITT population included all randomized participants whether or not they were assigned to the arm where the study treatment was administered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Venetoclax + Fulvestrant | Fulvestrant
Number analyzed (Participants) | 51 | 52
Months | 2.69 [1.94 to 3.71] | 1.94 [1.84 to 3.55]
Statistical Analysis 1: Comparison: Venetoclax + Fulvestrant vs Fulvestrant; Test type: Superiority; p = 0.7853, Regression, Cox — P-value is based on Stratified Analysis (Stratified by BCL2 status (High vs Low) and Lines of Therapy (2 vs 1)); Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.61 to 1.45]

3. Secondary Outcome: Objective Response (OR)
Description: OR was defined as CR or PR, in participants with measurable disease at baseline as determined by the investigator according to RECIST v1.1.
Time Frame: as for outcome 1
Population: The Baseline Measurable Disease Population represented all randomized participants with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Venetoclax + Fulvestrant | Fulvestrant
Number analyzed (Participants) | 51 | 51
Percentage of Participants | 3.9 [0.48 to 13.46] | 5.9 [1.23 to 16.24]
Statistical Analysis 1: Comparison: Venetoclax + Fulvestrant vs Fulvestrant; Test type: Superiority; p = 0.5978, Cochran-Mantel-Haenszel — P-value is based on Stratified Analysis (Stratified by BCL2 status (High vs Low) and Lines of Therapy (2 vs 1)); Risk Difference (RD) = -1.96, 95% CI 2-sided [-12.29 to 8.37]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first occurrence of a documented objective response to the time of the first documented disease progression (as determined by the investigator according to RECIST v1.1) or death from any cause, whichever occurs first.
Time Frame: Time from first occurrence of a documented objective response to the first documented disease progression or death from any cause, whichever occurs first, until 6 months after the last participant is enrolled in the study (up to approximately 23 months)
Population: Only participants with a documented objective response were analysed for this Outcome Measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Venetoclax + Fulvestrant | Fulvestrant
Number analyzed (Participants) | 2 | 3
Months | NA [NA to NA] — Insufficient number of participants meant that Median, Lower Limit and Upper Limit values could not be estimated. | 3.61 [1.94 to NA] — Insufficient number of participants meant that Upper Limit value could not be estimated.

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: Randomization to death from any cause, through till the end of the study (up to approximately 32 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Venetoclax + Fulvestrant | Fulvestrant
Number analyzed (Participants) | 51 | 52
Months | 19.71 [13.73 to NA] — Data for upper limit of CI was not estimable due to fewer number of participants with events. | NA [20.93 to NA] — Data for median and upper limit of CI was not estimable due to fewer number of participants with events
Statistical Analysis 1: Comparison: Venetoclax + Fulvestrant vs Fulvestrant; Test type: Superiority; p = 0.0403, Log Rank — P-value is based on Stratified Analysis (Stratified by BCL2 status (High vs Low) and Lines of Therapy (2 vs 1)); Hazard Ratio (HR) = 1.87, 95% CI 2-sided [1.02 to 3.43] — Hazard ratios were estimated by Cox regression

6. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study were also considered as AEs.
Time Frame: Baseline up until 28 days after the last dose of study drug (venetoclax or fulvestrant, whichever is later) up to approximately 32 months
Population: Safety-evaluable population which included all participants who received any amount of any component of the investigational or non-investigational study treatments.
Measure: Number; unit: Percentage of Participants
Arm/Group | Venetoclax + Fulvestrant | Fulvestrant
Number analyzed (Participants) | 50 | 51
Percentage of Participants | 94.0 | 76.5

7. Secondary Outcome: Plasma Concentrations of Venetoclax
Time Frame: Cycle 1 Day 1: 4 hours (hrs) post-dose; Cycle 2 Day 1: pre-dose (within 1 hr) and 2, 4, 6, 8 hrs post-dose; any time during visits up to study drug discontinuation/Early Termination (up to approximately 32 months)
Population: Pharmacokinetic (PK) evaluable population included all participants who received at least one dose of the study drugs (either venetoclax or fulvestrant) and had evaluable PK data. Number analyzed is the number of participants with data available for analyses at the given time-point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per Milliliters (μg/mL)
Groups:
- Venetoclax: Participants were administered Venetoclax 800mg orally QD and Fulvestrant 500mg IM on Day 1 and 15 of Cycle 1 and Day 1 of subsequent cycles (Cycle length = 28 days).
Arm/Group | Venetoclax
Number analyzed (Participants) | 47
Micrograms per Milliliters (μg/mL)
  Cycle 1 Day 1: 4 hrs post-dose | 1.78 (61.8)
  Cycle 2 Day 1: pre-dose: number analyzed (Participants) | 40
  Cycle 2 Day 1: pre-dose | 1.04 (85.4)
  Cycle 2 Day 1: 2 hrs post-dose: number analyzed (Participants) | 39
  Cycle 2 Day 1: 2 hrs post-dose | 1.45 (74.1)
  Cycle 2 Day 1: 4 hrs post-dose: number analyzed (Participants) | 40
  Cycle 2 Day 1: 4 hrs post-dose | 2.51 (57.2)
  Cycle 2 Day 1: 6 hrs post-dose: number analyzed (Participants) | 35
  Cycle 2 Day 1: 6 hrs post-dose | 3.32 (56.4)
  Cycle 2 Day 1: 8 hrs post-dose: number analyzed (Participants) | 28
  Cycle 2 Day 1: 8 hrs post-dose | 3.55 (57.8)
  Treatment discontinuation visit: number analyzed (Participants) | 21
  Treatment discontinuation visit | 0.0112 (NA) — Data for Geometric Coefficient of Variation was not reportable as more than one-third values were lower than reportable.

8. Secondary Outcome: Plasma Concentrations of Fulvestrant (in Presence of Venetoclax)
Time Frame: Cycle 2 Day 1: pre-dose (within 1 hr); Cycle 6 Day 1: pre-dose (within 1 hr); any time during visits up to study drug discontinuation/Early Termination (up to approximately 32 months)
Population: PK evaluable population included all participants who received at least one dose of the study drugs (either venetoclax or fulvestrant) and had evaluable PK data. Number analyzed is the number of participants with data available for analyses at the given time-point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Fulvestrant: Participants were administered Venetoclax 800mg orally QD and Fulvestrant 500mg IM on Day 1 and 15 of Cycle 1 and Day 1 of subsequent cycles (Cycle length = 28 days)
Arm/Group | Fulvestrant
Number analyzed (Participants) | 42
μg/mL
  Cycle 2 Day 1: pre-dose | 0.0129 (37.1)
  Cycle 6 Day 1: pre-dose: number analyzed (Participants) | 7
  Cycle 6 Day 1: pre-dose | 0.0145 (31.8)
  Treatment discontinuation visit: number analyzed (Participants) | 28
  Treatment discontinuation visit | 0.00985 (29.1)

9. Secondary Outcome: Plasma Concentrations of Fulvestrant (in Absence of Venetoclax)
Time Frame: Cycle 2 Day 1: pre-dose (within 1 hr); any time during visits up to study drug discontinuation/Early Termination (up to approximately 32 months)
Population: PK evaluable population included all participants who received at least one dose of the study drugs (either venetoclax or fulvestrant) and had evaluable PK data. Number of participants analyzed is the number of participants analyzed for this outcome measure. Number analyzed is the number of participants with data available for analyses at the given time-point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Fulvestrant
Number analyzed (Participants) | 5
μg/mL
  Cycle 2 Day 1: pre-dose | 0.0103 (29.4)
  Treatment discontinuation visit: number analyzed (Participants) | 1
  Treatment discontinuation visit | 0.0139 (NA) — Data for Geometric Coefficient of Variation was not estimable due to lower number of participants at given timepoint.

ADVERSE EVENTS:
Time Frame: Baseline up until 28 days after the last dose of study drug (venetoclax or fulvestrant, whichever is later) up to approximately 32 months.
Description: The 1 additional death in the Venetoclax + Fulvestrant arm compared to in the Participant Flow section, relates to a participant who had withdrawn consent from the study and later died. Their death was reported in public records (reported as a post study reporting death).
  All-cause mortality is for ITT population and serious and other AEs are reported for safety population.
Arm/Group | Venetoclax + Fulvestrant | Fulvestrant
All-Cause Mortality (participants affected / at risk) | 26/51 | 18/52
Serious Adverse Events (participants affected / at risk) | 4/50 | 2/51
Other Adverse Events (participants affected / at risk) | 45/50 | 34/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax + Fulvestrant (N=50) | Fulvestrant (N=51)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax + Fulvestrant (N=50) | Fulvestrant (N=51)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 8 (11) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 28 (39) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 32 (40) | 9 (10)
Vomiting (Gastrointestinal disorders) | 15 (23) | 1 (1)
Chest pain (General disorders) | 4 (4) | 0 (0)
Fatigue (General disorders) | 18 (20) | 9 (9)
Injection site reaction (General disorders) | 11 (15) | 15 (21)
Oedema peripheral (General disorders) | 4 (6) | 1 (2)
Hepatic pain (Hepatobiliary disorders) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Injection related reaction (Injury, poisoning and procedural complications) | 4 (6) | 5 (5)
Alanine aminotransferase increased (Investigations) | 2 (2) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 4 (4)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 2 (2)
Weight decreased (Investigations) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (2)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 7 (8) | 8 (8)
Insomnia (Psychiatric disorders) | 8 (8) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 9 (9)

LIMITATIONS AND CAVEATS:
The study was terminated due to Sponsor's decision and there were no safety concerns. Primary and secondary efficacy endpoints have been updated to report 95% confidence interval (CI) for Clinical Benefit estimate and 95% CI for the Cox proportional hazards model for PFS, following reporting conventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT03584009/Prot_SAP_001.pdf